CLINICAL TRIAL: NCT00232258
Title: Nolpitantium Besylate in Patients With Mild to Moderate Ulcerative Colitis, a Double-Blind, Placebo Controlled Efficacy and Safety, 8 Week Study
Brief Title: Nolpitantium Besylate In Patients With Ulcerative Colitis a Double-Blind, Placebo Controlled Efficacy and Safety Study
Acronym: NICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI4553
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: NK1 Antagonist; Inflammatory Bowel Disease; Mesalamine
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — SR 140333

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Nolpitantium besylate

SUMMARY:
To evaluate the safety and efficacy on clinical symptoms, mucosal histology and endoscopic mucosal appearance of two doses of SR140333B against placebo in patients with mild to moderate ulcerative colitis resistant to treatment with 5-ASA.

DETAILED DESCRIPTION:
Patients with active mild to moderate ulcerative colitis that has not responded to a minimum of 4 weeks of 5-ASA will be randomized to receive single daily doses of either placebo, 600 mg SR140333B or 1800 mg of SR140333B for eight weeks. Patients will undergo baseline and end of study sigmoidoscopic assessments and complete daily symptom diaries during the study. Ulcerative colitis disease activity will be measured by both the overall and component subscores of the Mayo Disease Activity Index.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Ulcerative colitis of at least 6 months duration
* Patient's ulcerative colitis should remain active while taking 5-ASA or sulfasalazine for at least 4 week
* If taking corticosteroids, dose must be stable for at least 2 weeks prior to enrollment and not exceed 20 mg per day (prednisolone equivalent)

Exclusion Criteria:

* Crohn's disease
* Colonic dysplasia
* Stool culture positive for enteric pathogens
* Concurrent cancer or unstable medical condition
* Recent treatment with monoclonal antibody
* Recent introduction of thiazolidinedione
* Recent treatment with methotrexate or cyclosporine
* Recent treatment with an antibiotic prescribed for ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2005-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Clinical remission at 8 weeks defined as a clinical Mayo subscore </= 1

SECONDARY OUTCOMES:
Clinical response defined as at least 3 point reduction from baseline on Clinical Mayo Sub-score
Global change in overall Disease Activity Index
Abdominal pain score at 8 weeks
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Gert Van Assche, MD, Principal Investigator — Universitaire Ziekenhizen Leuven
Locations (14):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com